CLINICAL TRIAL: NCT05196659
Title: Developing and Testing a Collaborative Quality ImProvement (C-QIP) Initiative for Prevention of Cardiovascular Disease in India
Brief Title: Collaborative Quality Improvement (C-QIP) Study
Acronym: C-QIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation of India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RA1055
Record Dates: First submitted 2021-12-02; First posted 2022-01-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease; Ischemic Stroke; Heart Failure
MeSH Terms: conditions — Coronary Disease; Ischemic Stroke; Heart Failure

STUDY DESIGN:
Intervention Model Description: Individual randomized parallel-group feasibility trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL Group (No Intervention): * Regular current system of care
  * Treating physicians provided current cardiovascular disease management guidelines
  * Patients provided a leaflet (printed information) on healthy lifestyle
- INTERVENTION Group (Active Comparator): 1. Electronic Health Record-Decision Support Software (EHR-DSS):
     * Electronic patient health record storage
     * Management prompts to the clinical team (following algorithms)
     * Structured follow-up schedule with automatic reminders to patients, clinical team, and non-physician health worker
  2. Non-physician health worker-led continuity of care:
     - individually tailored follow-up and guidance regarding treatment adherence as well as help in resolving issues related to access, convenience, cost of care, and equity
  3. Text-message based reminders for a healthy lifestyle
  4. Patient diary containing visual assessment tool for adherence to medication (VITA) and reinforcement tool for lifestyle modification
  5. Quarterly audit and feedback to the clinical team
  Interventions: Behavioral: Integrated comprehensive cardiovascular disease management

INTERVENTIONS:
Behavioral: Integrated comprehensive cardiovascular disease management — 1. Electronic Health Record-Decision Support Software (EHR-DSS):
     * Electronic patient health record storage
     * Management prompts to the clinical team (following algorithms)
     * Structured follow-up schedule with automatic reminders to patients, clinical team, and non-physician health worker
  2. Non-physician health worker-led continuity of care:
     - individually tailored follow-up and guidance regarding treatment adherence as well as help in resolving issues related to access, convenience, cost of care, and equity
  3. Text-message based reminders for a healthy lifestyle
  4. Patient diary containing visual assessment tool for adherence to medication (VITA) and reinforcement tool for lifestyle modification
  5. Quarterly audit and feedback to the clinical team
  Arms: INTERVENTION Group

SUMMARY:
The overarching goal of this study is to develop, implement, and evaluate the effect of a collaborative quality improvement (C-QIP) intervention (consisting of non-physician health workers, text messages for a healthy lifestyle, and a clinical decision support system) on processes of care and clinical outcomes among individuals with previous cardiovascular disease in India.

DETAILED DESCRIPTION:
Specific objectives of this study are:

1. To describe current practices, context, challenges, and opportunities regarding chronic management of cardiovascular disease from the patient, caregiver, provider, and health administrator perspectives in India.
2. To assess the transferability of components of internationally successful multifaceted quality improvement strategies and chronic care models to the Indian healthcare context.
3. To conduct a pilot study to assess the acceptability, feasibility, and implementation fidelity of the C-QIP strategy among individuals with cardiovascular disease attending out-patient clinics in India.
4. Among individuals with cardiovascular disease, evaluate the effect of C-QIP strategy on processes of care and clinical outcomes, health-related quality of life, and costs at 1 year compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

Participants should be:

* age ≥18 years, both sexes
* confirmed diagnosis of cardiovascular disease (ischemic heart disease, stroke, or heart failure irrespective of ejection fraction)
* able to provide written informed consent.

Exclusion Criteria:

* pregnant women
* those with any serious or uncontrolled medical condition (e.g., cancer) that may restrict the patient to come for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Implementation outcomes | at the end of study (maximum follow-up duration 24 months).
  Using mixed methods evaluation involving quantitative survey and in-depth interviews with the providers and patients, the primary outcome of this study is to assess the implementation outcomes such as the feasibility, and acceptability of the trial intervention defined as the extent to which providers and patients perceive the intervention strategy to be feasible to implement and useful/acceptable in their local health care setting.
Prescription of evidence based medicines | at the end of study (maximum follow-up duration 24 months).
  Through patient chart review, the study will assess the proportion of intervention arm versus control group participant's receiving evidence based medicines for cardiovascular disease management.
Adherence to prescribed therapy | at the end of study (maximum follow-up duration 24 months).
  Using validated questionnaire for medication adherence, the study will assess patient's compliance or adherence to prescribed therapy in the intervention group versus control group participants at the trial end.

SECONDARY OUTCOMES:
Change in blood pressure | at the end of study (maximum follow-up duration 24 months).
  Mean change in systolic and diastolic blood pressure between the intervention and control group participants at the trial end.
Change in low density lipoprotein cholesterol (LDLc) | at the end of study (maximum follow-up duration 24 months).
  Mean change in LDLc between the intervention and control group participants at the trial end.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Singh, PhD, Principal Investigator — Public Health Foundation of India
Locations (4):
- India (4):
  - SDM College of Medical Sciences and Hospital, Dharwad, Karnataka
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - GB Pant Hospital, New Delhi, New Delhi
  - Sir Ganga ram Hospital, New Delhi, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to other researchers upon reasonable request to the study PI.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be made available to other researchers after completion of the study and publication of primary results (Dec 2025).

REFERENCES:
- [Derived] Singh K, Roy A, Kondal D, Nikhare K, Gandral M, Patil SG, Aithal K, Girish MP, Gupta M, Madan K, Sawhney J, Ali K, Jain M, Kushwaha S, Jindal D, Mendenhall E, Patel SA, Venkat Narayan KM, Tandon N, Huffman MD, Prabhakaran D. A Randomized Feasibility Trial of a Multicomponent Quality Improvement Strategy for Chronic Care of Cardiovascular Diseases: Findings from the C-QIP Trial in India. medRxiv [Preprint]. 2026 Jan 30:2026.01.28.26345028. doi: 10.64898/2026.01.28.26345028. PMID 41646739
- [Derived] Singh K, Nikhare K, Gandral M, Aithal K, Patil SG, Mp G, Gupta M, Madan K, Sawhney JPS, Ali K, Kondal D, Jindal D, Mendenhall E, Patel SA, Narayan KMV, Tandon N, Roy A, Huffman MD, Prabhakaran D. Rationale, Design and Baseline Characteristics of a Randomized Controlled Trial of a Cardiovascular Quality Improvement Strategy in India: The C-QIP Trial. Am Heart J. 2024 Oct;276:83-98. doi: 10.1016/j.ahj.2024.07.008. Epub 2024 Jul 20. PMID 39033994